CLINICAL TRIAL: NCT02453607
Title: The Impact of 6MP Metabolite Levels on Infliximab Pharmacokinetics and Anti-infliximab Antibodies in Crohn's Disease
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Ernest Seidman (Other)
Collaborators: University of Toronto (Other); University of Calgary (Other); University of Alberta (Other)
Responsible Party: Sponsor-Investigator, Ernest Seidman, Professor of Medicine & Pediatrics, McGill University Health Centre/Research Institute of the McGill University Health Centre
Organization: McGill University Health Centre/Research Institute of the McGill University Health Centre (Other)
Other Study IDs: 14-158-GEN
Record Dates: First submitted 2015-05-21; First posted 2015-05-25 (Estimated); Last update posted 2017-02-16 (Actual); Status verified 2017-02

CONDITIONS: Inflammatory Bowel Disease; Crohn's Disease
MeSH Terms: conditions — Inflammatory Bowel Diseases; Crohn Disease | interventions — Infliximab; 2-mercaptopurine; Azathioprine

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — We will be storing, de-identified, blood samples on site in the lab of Dr Ernest Seidman
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- CD Monotherapy: Crohn's disease treated with infliximab (monotherapy)
  Interventions: Drug: Infliximab
- CD Combo therapy: Crohn's disease treated with infliximab in combination with thiopurine (a 6MP metabolite) (combo therapy)
  Interventions: Drug: Infliximab; Drug: thiopurine

INTERVENTIONS:
Drug: Infliximab — Drug is prescribed by treating physician and is not a part of the study. This study is non-interventional. Patients, to be elgibile, are being prescribed either monotherapy inlfiximab or combo therapy infliximab with azathiopurine.
  Other Names: Remicade
Drug: thiopurine — Drug is prescribed by treating physician and is not a part of the study. This study is non-interventional. Patients, to be elgibile, are being prescribed either monotherapy inlfiximab or combo therapy infliximab with azathiopurine.
  Other Names: Imuran
  Groups: CD Combo therapy

SUMMARY:
In this research proposal, the investigators will focus on methods to optimize the therapeutic response to anti-TNF antibodies, by determining a correlation of 6-mp metabolite levels with IFX trough levels, anti-IFX antibody levels and clinical response. The study will also evaluate (in vitro) the possible impact of vitamin D on the interaction of IFX with dendritic cells in both healthy subjects and patients with Crohn's disease (proliferation, maturation, cytokine profile, apoptosis, gene expression).

DETAILED DESCRIPTION:
Despite the evidence for the beneficial effects of thiopurine/IFX combined therapy on both the prevention of the development of anti-IFX antibodies (ATI) and improved clinical outcomes, no study has employed the proven clinical usefulness of measuring 6- MP metabolite levels. We hypothesize that targeting the established threshold of 6-TGN levels (between 235-400), shown to result in superior clinical efficacy, would reduce the development of ATI and enhance trough IFX levels. It is also conceivable that excessive6TGN levels may increase the risk of adverse events such as infections and neoplasms such as lymphomas, the major drawbacks to combination therapy. If a significant correlation between 6-TGN levels and diminished risk of ATI development or higher trough serum IFX levels can be demonstrated, it will allow for an improved approach towards pharmacological monitoring of these patients with optimization of the long term response of CD patients on anti-TNF therapy.

Vitamin D possesses profound immunomodulatory effects, mediated primarily through the innate immune system. Low serum levels of vitamin D are associated with worse outcomes in CD. IFX was reported to have a significant impact on maturation and phenotype of dendritic cells (DC). Previous work from our laboratory demonstrated a significant effect of vitamin D on expression of NOD2 along with a profound effect onthe cytokine profile of DC exposed to PRR stimulation85. We hypothesize that vitamin Ddeficiency may be associated with a lower clinical response to anti-TNF therapy. IFX and vitamin D may have a synergistic effect in modulating the immune system in IBD via interactions through innate or adaptive mechanisms. We expect that vitamin D may enhance IFX-induced shift in the maturation pathway and cytokine profile of DC exposed to intestinal microbes through pattern recognition receptors (PRR). Demonstration of a synergistic effect of vitamin D with anti-TNF antibodies may have important clinical implications for the care of IBD patients, particularly in Canada where the prevalence of vitamin D deficiency is very high. Such an effect was demonstrated for lymphocytes but was never examined for the innate immune system, considered to have a profound role in the pathogenesis of CD. The data from this study may provide further justification for the need of monitoring vitamin D status in CD patients, and its supplementation as an additional therapeutic tool for optimizing response to anti-TNF in CD.

This is a prospective cross-sectional and longitudinal multicentre non-interventional study. The patients will be recruited at the following centers: McGill University Health Center, Mount Sinai Medical Centre, Toronto, Canada; University of Calgary, U Alberta, Edmonton. This study will recruit patients (18-70 yrs) with Crohn's disease who are starting treatment with infliximab or combo therapy of infliximab and azathiopurine. This study will look at therapeutic monitoring end points to evaluate the impact of drug level and antibodies on the clinical effectiveness of treatment (mono or combo therapy). .

ELIGIBILITY:
Inclusion Criteria:

* Patients with a diagnosis of CD ,
* age 18-70 years,
* who are treated with IFX (standard 5 mg/kg/q8 weeks maintenance dose) or IFX (standard maintenance dose)/thiopurine (stable dose for at least 3 months) combination for <12 months.-

Exclusion Criteria:

* Age< 18 years;
* Patients treated with IFX at non-standard doses;
* diagnosis of ulcerative colitis, pouchitis, indeterminate colitis or Crohn's disease involving the upper GI tract or perianal disease without involvement of small bowel or colon;
* concomitant therapy with cyclosporine, methotrexate or other immunosuppressant other than thiopurine and IFX, treatment with IFX or IFX/thiopurine combination for > 12 months;
* pregnancy

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Patients with a diagnosis of CD ,age 18-70 years, who are treated with IFX (standard 5 mg/kg/q8 weeks maintenance dose) or IFX (standard maintenance dose)/thiopurine (stable dose for at least 3 months) combination for <12 months.
Sampling Method: Probability Sample
Enrollment: 225 (Estimated)
Dates: Start 2014-11-17 (Actual); Primary Completion 2019-06-30 (Estimated); Study Completion 2020-06-30 (Estimated)

PRIMARY OUTCOMES:
Correlation of 6-TGN serum levels with IFX serum trough levels | 52 weeks
  Evaluate the correlation of 6-TGN serum levels with IFX serum trough levels , prevalence of ATI and clinical response treatment in CD patients treated with a combination of IFX and a thiopurine.

SECONDARY OUTCOMES:
Evaluation of 6-TGN serum levels and IFX trough levels | 52 weeks
  Evaluate the correlation of 6-TGN serum levels at the initial visit (week 14 or visit 1) with IFX serum trough levels, prevalence of ATI and clinical response at week 52.
6 TGN levels and dose escalation or disconinuation of IFX | 52 plus 6 months for data calculation
  Determine the correlation of 6-TGN levels with need for dose escalation and discontinuation of IFX for the duration of the study.
Vitamin D levels and efficacy of anti-TNF therapy | duration of study and 1 additional year for data analysis
  Evaluate the correlation of vitamin D levels (sufficient, insufficient, deficient) on the efficacy of anti-TNF therapy in patients with Crohn's disease.
Vitamin D status and effect on ATI levels | duration of study and 1 additional year for data analysis
  Determine the correlation between vitamin D status with trough IFX levels and the prevalence of ATI.

CONTACTS AND LOCATIONS:
Overall Officials: Ernest Seidman, MDCM, Principal Investigator — McGill University Health Centre/Research Institute of the McGill University Health Centre
Locations (1):
- Montreal General Hospital, Montreal, Quebec, Canada

IPD SHARING:
Plan to Share IPD: No